CLINICAL TRIAL: NCT01039155
Title: A Phase 1 Study of CTEP 5-Azacytidine in Combination With Oxaliplatin in Patients With Advanced Cancers Relapsed or Refractory or Refractory to Any Platinum Therapy
Brief Title: Azacitidine and Oxaliplatin In Treating Patients With Advanced Cancers Relapsed or Refractory to Any Platinum Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02909; NCI-2012-02909 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 662917; 2008-0277; 2008-0277 (Other: M D Anderson Cancer Center); 8321 (Other: CTEP); P30CA016672 (NIH); U01CA062461 (NIH)
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-05

CONDITIONS: Adult Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Azacitidine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (azacitidine, oxaliplatin) (Experimental): Patients receive azacitidine IV over 15-30 minutes on days 1-5 and oxaliplatin IV over 2 hours on days 2-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Other: Laboratory Biomarker Analysis; Drug: Oxaliplatin; Other: Pharmacological Study

INTERVENTIONS:
Drug: Azacitidine — Given IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I clinical trial studies the side effects and the best dose of azacitidine and oxaliplatin in treating patients with advanced cancers that do not respond to treatment or have returned after any platinum therapy. Azacitidine is designed to activate (turn on) certain genes in cancer cells whose job is to fight tumors. Oxaliplatin is designed to block the growth and spread of new cancer cells, eventually destroying them, by damaging their deoxyribonucleic acid (DNA). Giving azacitidine with oxaliplatin may kill more cancer cells and may also reverse resistance to platinum-based drugs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of 5-azacytidine (azacitidine) and oxaliplatin combination regimen in patients with advanced solid tumors or lymphomas relapsed or refractory to any platinum compound.

II. To define 5-azacytidine and oxaliplatin pharmacokinetics.

SECONDARY OBJECTIVES:

I. For patients treated in the expansion phase of this study: (a) to assess copper transport protein (CTR1) score; (b) to assess changes in global DNA methylation; and (c) to measure changes in oxaliplatin levels in tumor biopsies between pretreatment and day 12 of the first cycle of 5-azacytidine plus oxaliplatin therapy.

II. To correlate results of the pharmacokinetic studies of 5-azacytidine and oxaliplatin with changes in CTR1, changes in global DNA methylation and changes in oxaliplatin levels in tissue biopsies of patients treated in the expansion phase of this study.

OUTLINE: This is a dose-escalation study.

Patients receive azacitidine IV over 15-30 minutes on days 1-5 and oxaliplatin IV over 2 hours on days 2-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy (solid tumor or lymphoma) that is metastatic or unresectable and for which standard curative or palliative measures are not expected to increase survival by at least 3 months
* Patients must have an advanced cancer relapsed or refractory to any platinum compound; platinum-refractory disease is defined as disease that does not respond to a platinum compound-containing regimen or that recurs after treatment with a platinum compound-containing regimen
* Patients must have had >= 1 prior chemotherapy regimen; there is no maximum allowable number of prior regimens, provided all other eligibility criteria are met
* Patients must be >= 6 weeks beyond treatment with a nitrosourea or mitomycin-C, >= 4 weeks beyond other chemotherapy or radiotherapy, and must have recovered to =< grade 1 toxicity for any treatment-limiting toxicity of prior therapy; (exception: patients may have received palliative low-dose radiotherapy to the limbs 1-4 weeks before this therapy, provided pelvis, ribs, sternum, scapulae, vertebrae, or skull were not included in the radiotherapy field)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 4,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< 1.0 mg/dL
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 3 X institutional upper limit of normal
* Creatinine (serum) =< 2.0 mg/dL
* International normalized ratio (INR) of less than or equal to 1.75 per institutional guideline
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients must have the ability to understand and the willingness to sign a written informed consent document, including consent for the required tumor biopsy (in the expansion phase), blood, and pharmacokinetics studies
* Tumor should be accessible for repeat biopsy if in the expansion phase; biopsies will be performed in the expansion phase; the expansion cohort will be between 10 and 20 patients
* Patients must have expected survival of at least 3 months

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered to =< grade 1 treatment-limiting toxicity levels for adverse events due to agents administered more than 4 weeks earlier; (exception: patients may have received palliative low dose radiotherapy to the limbs 1-4 weeks before this therapy, provided pelvis, ribs, sternum, scapulae, vertebrae, or skull were not included in the radiotherapy field)
* Patients may not be receiving any other concurrent investigational agents
* Patients must not have a history of allergic reactions attributed to 5-azacytidine, oxaliplatin, or compounds with a similar composition
* Patients must not have oxaliplatin intolerance
* Patients must not have uncontrolled intercurrent illness, including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, potentially life-threatening cardiac arrhythmia, and psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with 5-azacytidine
* Patients known to be human immunodeficiency virus (HIV)-positive and receiving anti-retroviral therapy must have both a minimum of 350 CD4+ cells/mm^3 and no history of acquired immunodeficiency syndrome (AIDS) defining conditions except for lymphoma
* Patients who have had surgery within 2 weeks prior to entering the study are not eligible
* Patients who have been removed from prior platinum-containing therapy due to platinum-compound cumulative toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-12; Primary Completion 2012-09 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
MTD graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 28 days

SECONDARY OUTCOMES:
Changes in concentration of oxaliplatin | Baseline to day 12
Changes in DNA methylation | Baseline to day 12
Changes in the CTR1 score | Baseline to day 28
Pharmacokinetic parameters of azacitidine and oxaliplatin | Days 1 and 5 of course 1 (azacitidine) and day 2 of course 1 (oxaliplatin)
  Compartmental and non-compartmental modeling will be used to derive pharmacokinetic parameters, including maximum concentration (Cmax), time to maximum plasma concentration (Tmax), area under the curve (AUC), t ½ alpha (a), t ½ beta (B), volume of distribution (Vd), and clearance.

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia-Maria Tsimberidou, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States